CLINICAL TRIAL: NCT03096431
Title: Does Cognitive Rehabilitation and Physical Activity Impact Executive Functioning Following Radiation Therapy for Cerebral Metastases? A Pilot Study
Brief Title: Impact of Cognitive Rehab and Physical Activity on Cognition in Patients With Metastatic Brain Tumors Undergoing RT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution: Will not continue study.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MCC-16-13082; HM20007924 (Other: IRB)
Record Dates: First submitted 2017-03-23; First posted 2017-03-30 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Brain Tumor; Cerebral Metastases
Keywords: whole-brain radiation therapy; sterotactic radiosurgery; cognitive rehabilitation; physical activity
MeSH Terms: conditions — Brain Neoplasms; Motor Activity | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: All participants will be blinded to the study design and will be randomized into one of three treatment arms. Research assistant is blinded to both the study design and to which arm the participants are randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Physical activity intervention (Active Comparator): Undergo baseline testing of physical (lower body strength, endurance) and cognitive (executive functioning) abilities. 14 days (± 2 days) following WBRT/SRS: all arms undergo testing of physical (lower body strength, endurance) and cognitive (executive functioning) abilities. Arm 1: intervention of physical activity begins. 60 days (± 5 days) post testing after WBRT/SRS: all arms undergo final testing of physical (lower body strength, endurance) and cognitive (executive functioning) abilities.
  Interventions: Behavioral: Physical Activity
- Arm 2:Physical activity and cognitive intervention (Active Comparator): Undergo baseline testing of physical (lower body strength, endurance) and cognitive (executive functioning) abilities. 14 days (± 2 days) following WBRT/SRS: all arms undergo testing of physical (lower body strength, endurance) and cognitive (executive functioning) abilities. Arm 2: intervention of both cognitive rehabilitation and physical activity begins. 60 days (± 5 days) post testing after WBRT/SRS: all arms undergo final testing of physical (lower body strength, endurance) and cognitive (executive functioning) abilities.
  Interventions: Behavioral: Physical Activity; Behavioral: Cognitive rehabilitation
- Arm 3: Cognitive and begin physical activity intervention (Active Comparator): Undergo baseline testing of physical (lower body strength, endurance) and cognitive (executive functioning) abilities. Arm 3: Intervention of cognitive rehabilitation begins prior to and is concurrent with WBRT/SRS treatment. 14 days (± 2 days) following WBRT/SRS: all arms undergo testing of physical (lower body strength, endurance) and cognitive (executive functioning) abilities. Arm 3: continue intervention of cognitive rehabilitation; add intervention of physical activity. 60 days (± 5 days) post testing after WBRT/SRS: all arms undergo final testing of physical (lower body strength, endurance) and cognitive (executive functioning) abilities.
  Interventions: Behavioral: Physical Activity; Behavioral: Cognitive rehabilitation

INTERVENTIONS:
Behavioral: Physical Activity — * Self-exercise: number of steps per day, per fitness tracker; self-report of daily activity.
  * One-to-one intervention: 30 minute sessions with licensed therapist to include warm-up, generalized strengthening, stretching.
  Other Names: PA
Behavioral: Cognitive rehabilitation — One-to-one intervention: 45 minutes sessions with licensed therapist to include graded cognitive tasks designed to improve executive functioning with focus on both restorative and compensatory approaches.
  Other Names: CR; Cognitive retraining
  Arms: Arm 2:Physical activity and cognitive intervention; Arm 3: Cognitive and begin physical activity intervention

SUMMARY:
To determine the feasibility of processes and instruments with an overarching purpose to guide the design of a larger study. To determine the feasibility of individuals with metastatic brain tumor(s) to engage in physical activity(PA) and cognitive rehabilitation (CR) as in an outpatient therapy setting.

DETAILED DESCRIPTION:
Rolling recruitment for the study. Participants will be randomized into one of three treatment arms. All treatment arms will undergo physical & cognitive testing prior to whole-brain radiation therapy (WBRT)/stereotactic radiosurgery (SRS). Arm 3 will receive cognitive rehabilitation intervention sessions prior to, and concurrent with, WBRT/SRS. Approximately 14 days following WBRT/SRS: all arms will undergo physical and cognitive testing, and: Arm 1 will begin physical activity intervention. Arm 2 will begin physical activity intervention and cognitive intervention. Arm 3 will continue with cognitive intervention and begin physical activity intervention. All Arms will undergo physical and cognitive testing approximately 2.5 months post WBRT/SRS.

ELIGIBILITY:
Inclusion Criteria:

* A potential subject must meet all of the following inclusion criteria to be eligible to participate in the study:
* Ability to understand and the willingness to provide written informed consent
* 18 years of age and older
* Diagnosed with one or more metastatic brain tumor(s)
* Medical treatment plan includes whole-brain radiation therapy and / or sterotactic radiosurgery

Exclusion Criteria:

* A potential subject who meets any of the following exclusion criteria is ineligible to participate in the study.
* Diagnosis of dementia or unable to grant their own informed consent
* Prisoner or patient in custody
* Patient on psychiatric hold
* Physically unable to participate in the study
* The opinion of the treating physician determines it is not medically safe to participate in the study
* Pre-registration screen of cognition is "severe" or lower.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
Recruitment percentage of eligible subjects. | 18.5 months
  Recruitment: success defined as enrollment rate of 19% of eligible subjects.
Retention percentage of participants at end-of-study. | 18.5 months
  Retention: success defined as retention rate above 56% at end-of-study.
Non-attendance rates of participants. instructions. | 18.5 months
  Participant missed or cancelled therapy sessions less than 15% of time.
Lengths of sessions completed. | 18.5 months
  Participant completed full scheduled minutes per session ≥ 80% of time.
Percentage of completion of Physical Activity intervention tasks. | 18.5 months
  Participant completed ≥ 80% of PA interventions (required < 20% rest period during or between tasks).
Percentage of Cognitive Therapy intervention tasks. | 18.5 months
  Participant completed ≥ 80% of CR interventions (required < 20% rest period during or between tasks).

SECONDARY OUTCOMES:
Change in cognitive abilities. | 18.5 months
  Composite score post-CR intervention, minus the composite score at baseline. Scores of zero indicates maintained cognition. Positive scores indicate improved cognition. Negative scores indicate declined cognition. Composite scores derived from the following four standardized tests:
  * The Stroop Color Word Test (SCWT) is a 3-part measure that tests the executive function area of attention.
  * The Trail Making Test (TMT) is a 2-part measure that tests the executive function area of complex attention.
  * The Rey Auditory Verbal Learning Test (AVLT) is a 6-part measure that tests the executive function area of memory.
  * The Clock Drawing Test (CDT) is a single measure that tests the executive function area of visuospatial relationships and praxis.
Change in physical abilities. | 18.5 months
  Composite scores post intervention minus scores at baseline. Scores of zero indicate maintained physical abilities. Positive scores indicate improved physical abilities. Negative scores indicate declined physical abilities. Composite scores derived from the following two standardized tests:
  * The Timed Up and Go (TUG) is a single measure that tests mobility, balance, and walking ability.
  * The 30-second Chair Stand Test (30sCST) is a single measure that tests functional lower body strength.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne F. Taylor, PhD, MBA, OTR/L, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States